CLINICAL TRIAL: NCT02880111
Title: Comparison of Rates DMBT1 ( Glycoprotein) in Sputum of CF Patients Colonized Patients Between Chronic and Non-chronic Patients Colonized With Pseudomonas Aeruginosa
Brief Title: Rates DMBT1 ( Glycoprotein) in Sputum of CF Patients With Pseudomonas Aeruginosa
Acronym: DMBT1
Status: Terminated | Type: Observational
Why Stopped: only one patient was included
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2012_44; 2014-A00259-38 (Other: ID-RCB number, ANSM); PHRCI-2012 (Other: PHRC number, DGOS)
Record Dates: First submitted 2016-08-23; First posted 2016-08-26 (Estimated); Last update posted 2022-10-18 (Actual); Status verified 2020-08

CONDITIONS: Malignant Brain Tumor
Keywords: Malignant Brain Tumor; patient sputum
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group 1: CF patients with Pseudomonas aeruginosa chronic colonization.
- group 2: CF patients without a Pseudomonas aeruginosa chronic colonization.

SUMMARY:
Rates of DMBT1 (Glycoprotein like) in Sputum of CF Patients with or without may be different according to their Pseudomonas Aeruginosa chronic colonization status. The aim of this study is to compare rates of DMBT1 (Glycoprotein like) in Sputum of CF patients with or without a Pseudomonas Aeruginosa chronic colonization.

DETAILED DESCRIPTION:
Rates of DMBT1 (Deleted in Malignant Brain Tumor 1) will be compared between 2 groups of 30 CF patients : group 1 : with Pseudomonas Aeruginosa chronic colonization and group 2 30 CF patients without Pseudomonas Aeruginosa chronic colonization.

ELIGIBILITY:
Inclusion Criteria:

* CF patient 6 years
* Availability of sputum
* Signed Informed consent

Exclusion Criteria:

* Cardiac insufficiency
* Anti-inflammatory drugs on going
* Oral corticosteroid therapy
* Inhaled corticosteroids during the two weeks before inclusion,
* Patient awaiting lung transplantation
* Patient with a past history of heart/lung transplantation
* Patient with a sputum examination positive for : atypical mycobacteria, Burkholderia cepacia, Stenotrophomonas maltophilia,
* Patient chronically colonized with multiresistant Pseudomonas aeruginosa
* Orkambi© or Kalydeco© therapy
* Change of the CF treatment during the last 4 weeks +/- 2 days before inclusion : corticosteroid, pancreatic extracts, antisecretory drugs...

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: CF Patients with or without Pseudomonas aeruginosa chronic colonization status aged 6 years.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2016-03-23 (Actual); Primary Completion 2022-03 (Actual); Study Completion 2022-03 (Actual)

PRIMARY OUTCOMES:
measure glycoprotein-like DMBT1 by Elisa | at 1 months
  DMBT1 in mg DMBT1 / mg of total protein measured by BCA (BiCinchoninic acid Assay) present in each sputum

SECONDARY OUTCOMES:
measure MUC5B by Elisa | at 1 months
  MUCB in mg / mg of total protein measured by BCA present in each sputum

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Turck, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Jeanne de Flandre - CHRU de Lille, Lille, France

IPD SHARING:
Plan to Share IPD: No